CLINICAL TRIAL: NCT05123430
Title: Hemodynamic Estimation Per Procedure of the Result of the MitraClip Technique: Interest of the Ratio of Mean Arterial Pressure (MAP) to Pressure of the Mean Left Atrium (POG)
Brief Title: Hemodynamic Estimation of the Result of the MitraClip Technique: Interest of the Ratio of Mean Arterial Pressure (MAP) to Pressure of the Mean Left Atrium (POG) (MitraPOG)
Acronym: MitraPOG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-A02328-31
Record Dates: First submitted 2021-11-09; First posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Mitral Insufficiency; Mitraclip
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MitraClip operated patients suffering from serious mitral insufficiency (Experimental)
  Interventions: Procedure: Monitoring of the pressure of the middle left atrium

INTERVENTIONS:
Procedure: Monitoring of the pressure of the middle left atrium — During the MitraClip surgery, additional catheter is installed in order to monitoring the ppressure of the middle left atrium

SUMMARY:
this research is based on the hypothesis that the measurement of the ratio of mean arterial pressure to mean left atrium pressure and of its evolution during the procedure, would make it possible to assess the immediate success of the procedure by supplementing the results of the ultrasound.

The main objective of this research is to define the percentage of improvement in the mean arterial pressure / mean left atrium pressure ratio at the end of the procedure to validate the success of the MitraClip procedure.

ELIGIBILITY:
Inclusion Criteria:

* Woman or man over 18 years old
* Patient with symptomatic mitral leakage (grade 3+ or 4+) at high surgical risk defined as:

  * Age ≥ 75 years and an STS score ≥ 6%, or, according to MVARC, at least 1 fragility index or at least 1 organ fragility criterion or at least 1 operative risk criterion. MVARC recommendations are defined in the appendix.
  * Age <75 years and an STS score> 8%, or, according to MVARC, at least 1 fragility index or at least 1 organ fragility criterion or at least 1 operative risk criterion. MVARC recommendations are defined in the appendix.
  * Patient rejected for surgery.
* Patient with a life expectancy of over 1 year.
* Patient affiliated or beneficiary of a social security scheme.
* Patient having been informed and having signed a written consent.

Exclusion Criteria:

* Patient with unfavorable ultrasound parameters (for example: patient with insufficient mitral surface).
* Patient with recent or active infection.
* Patient with a contraindication to the transseptal puncture.
* Patient with valve anatomy incompatible with the placement of the device.
* Patient with an anomaly of the tricuspid valve justifying a surgical intervention.
* Patient who has had a percutaneous cardiovascular procedure within the previous 30 days.
* Patient who had heart surgery in the previous 30 days.
* Patient with a history of surgery on the mitral valve.
* Patient having had a stroke in the previous 30 days.
* Patient participating in another clinical study.
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision.
* Pregnant, breastfeeding or parturient woman.
* Patient hospitalized without consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-03-23 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2022-03-23 (Estimated)

PRIMARY OUTCOMES:
Percentage improvement in the mean arterial pressure / mean left atrium pressure ratio measured at the end of the procedure. | 6 months
  The percentage of improvement is defined by the value (B-A) / A * 100, with A = mean arterial pressure / mean left atrium pressure ratio at the start of the procedure and B = mean left atrium pressure / mean arterial pressure ratio at the end of the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Médipôle Hôpital Privé, Villeurbanne, France